CLINICAL TRIAL: NCT06563232
Title: 22G-Adapt Needle Biopsy Versus Fine-needle Aspiration in Endoscopic Ultrasound-guided Sampling of Solid Lesions: a Randomized Controlled Study
Brief Title: 22G-Adapt Needle Biopsy Versus Fine-needle Aspiration in Endoscopic Ultrasound-guided Sampling of Solid Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Peking Union Medical College Hospital (Other); Fudan University (Other); Qilu Hospital of Shandong University (Other); Chongqing University Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Bin Cheng, prof., Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FNA vs Adapt FNB
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Neoplasms; Mediastinal Neoplasms; Abdominal Neoplasm, Excluding Pancreas Neoplasm
Keywords: endoscopic ultrasound; fine-needle aspiration; fine-needle biopsy
MeSH Terms: conditions — Pancreatic Neoplasms; Mediastinal Neoplasms; Abdominal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FNA group (Experimental): FNA needles adopted to acquire lesion tissues
  Interventions: Device: FNA group
- Adapt FNB group (Experimental): Adapt FNB needles adopted to acquire lesion tissues
  Interventions: Device: Adapt FNB group

INTERVENTIONS:
Device: FNA group — Fine-needle-aspiration (22G EchoTip Ultra Echo-3-22)
  Arms: FNA group
Device: Adapt FNB group — Fine-needle-biopsy (22G Adapt Aspiration)
  Arms: Adapt FNB group

SUMMARY:
The investigators conduct a multicenter randomized controlled study to evaluate the diagnostic value and safety of 22G Adapt Aspiration puncture needle for histopathology of solid lesions.

DETAILED DESCRIPTION:
The study subjects are divided into two groups: the EUS-FNA(22G EchoTip Ultra needles) Group and EUS-FNB group(22 Adapt Aspiration).Take the malignant occupying lesion diagnosis accuracy as the research major indicator to compare the EUS-FNB group and EUS-FNA group as optimal efficiency test. Take the class I error a=0.05, class II error β=0.15, power=0.85. Suppose the malignancy diagnosis accuracy is 82%, while that of FNB is 91%. The two trial groups be randomly allocated in 1:1, suppose the malignancy cases take 85% of the whole case, and considering the shedding factors , extra 20% cases should be included. So the estimated cases numbers is 328 cases for EUS-FNB group and 328 cases for EUS-FNA group, totally 656 cases in this trial.

Done by professional statistical people with randomized block grouping method and SAS 9.4 statistical software to generate randomized serial number（001-656）for the two groups in 1:1 manner. The serial numbers are the randomized grouping numbers for the trial patients, block capacity is 116, totally 41 randomized block. The randomized grouping will be generated in duplicate copies and sealed. One copy send to trial centers for patient allocating, and the another copy be saved by the trial applicant unit. Every trail centers will be responsible for the screening of qualified patients, rank them in visit time to get the randomized grouping number so as to determine them goes to the EUS-FNA or EUS-FNB.The research people and patients in all trial centers should not know the the randomized grouping number and relevant groups. The group name will be sealed under scratch card. Every trial patients will get a unique randomized number, and it will not change through out the whole trial.

Use the inclusion and exclusion criteria to observe the patients and do relative inspections, and confirm if the patients qualified or not to the trial. Record the result of last time test before the treatment. Although it is better to get the informed consent before doing all kinds of observation and tests, if for some reason, the medical imaging examination has completed, as long as the imaging examination was done within 3 weeks before the needle biopsy, it can still be collect as baseline data (imaging examination can be done at other hospitals, but the trial center should issue a new evaluation report 1 week before the patient join the trial group); other lab test items done at 2 weeks before the needle biopsy can still be collect as baseline data for pre-research use, but these tests should be done at the trail center hospital so as to guarantee the data trace ability.

The investigators will do the needle passes for 3 times for all of them:the 1 needle passes with Slow-Pull and the 2-3 needle passes with wide suction. If no core tissues obtained or the operator/onsite pathologist determine insufficient specimen after the operations above, then remedy procedures will be done, the operator use proper puncture method to continue the remedy biopsy. After the first round of needle biopsy, if the trial patient cannot be diagnosed, by getting the agreement of the patient, the patient will be cross-over to another trial group and do needle biopsy again on the same lesion 1 week later with the method mentioned above. Without knowing the needle biopsy type, the cytologist and pathologist evaluate the specimen quality and make diagnosis. Every specimen will be independently evaluated and diagnosed by 2 experts. If the 2 experts have different judgments, then these two experts discuss together and make the final diagnose discussion. If the same sample has 2 or more cytology smear slides, than take the highest score slide as the result. Follow up (outpatient follow up or telephone follow up) the patients at 1 week, 12 weeks and 36 weeks after the needle biopsy and collect the patients clinical data and confirm their final diagnosis.

During the trial, if severe adverse event occurs, the trialed center must take immediate actions necessary to guarantee the trialed patients' safety. Once severe adverse event occurs, the researchers should inform the trial applicant and the trail center's ethics committee within 24 hours after the researchers gets to know the adverse event. And the researchers should also fax the report to State Food and Drug Administration of China and the local provincial food and drug administration. After receiving the report, the applicant should inform other clinical trial centers within 24 hours. All the severe adverse events should be filed at group leader medical center and other trial centers.

CRF(Case Report Form ) will be filled by the researchers, every involved patient must have the CRF(Case Report Form ) filled. This will be audited by clinical monitor and handed over to data administrator to input and manage data, the first copy will be kept by the applicant, the second copy will go to the trial center, and the third copy will be kept by the trail researchers.The data input and management will be taken care by specially assigned person. In order to guarantee the data accuracy, data input will be done twice by two independent data administrators, by computerized and manual verifying, hand over the data to statistical experts to do blind check and statistic analyzing.For the questions and doubts within the case report form, the data administrator make DRQ and via the clinical monitor asking the researchers. The researchers will answer and feed back as soon as possible. According to the researchers answer, data administrator will do the data modifying, confirming or inputting, and when necessary send out DRQ again.After blind audition and confirming that the established data base is correct, major researchers, applicant and the statistic analyzing people lock the data. The locked data will not be changed, and the data base will be handed over to statistical analyzer to do the statistic analyze according to the statistic analyzing plan. Problems found after data locking can be modified during the statistic analyzing procedure.This will be done by specialized statistic analyzing people according to the predetermined statistic analyzing plan. The statistic analyze will be carried out according to intention principle confirmed full analysis set and per-protocol set principle. After completing the statistic analyzing, the statistic analyzer issue the statistic analysis report and send this to major researchers to write the study report.

Statistic analyzing plan:⑴ General principle:① all the statistic tests are use the two-tailed-test method, P<0.05 will be thought as the tested difference is statistical significance. ② the quantitative indicator description will calculate the Mean and Standard deviation. The classification indicator description will describe the cases and percentage of all types of cases. ⑵ Statistic analyzing method:① for the measurement data, compare it with the baseline value at selection period, use paired t-test or symbol rank sum test to compare with the before-after-difference within the group.② for the counting data, use x2 test or Fisher's exact test method to compare the groups. ⑶ Shedding analysis:Comparison of groups'total shedding rates and the shedding rates caused by adverse events will use x2 test or Fisher's exact test method. ⑷ The baseline value's equilibrium analysis: Use group t test or x2 test to compare the demography info and vital signs, disease history, and basic treatment and other indicators of baseline value, so as to measure the balance of the groups. The baseline evaluation will be done on FAS（full analysis set) and PPs(per-protocol set). ⑸ Effectiveness analysis:The major indicator of effectiveness analysis is the diagnostic accuracy on malignant disease, and the indicators of second effectiveness include the percentage of Grade A specimen and complications rate etc. while the two groups rate and the Youden index comparison will use approximate normal Z test or use central effect x2 test.(6) Safety analysis:Use x2 test or Fisher's exact test to compare the adverse event/adverse reaction (include biopsy complications) rates between the groups. And use table to describe the adverse events during this trial project; the lab test results before and after the trial, the normal/abnormal changing condition and the relationship with this trial research when abnormal changes happened.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old and under 85 years old;
* Imaging examinations (MRI, CT, B-ultrasound) reveal the presence of solid masses (with a diameter > 1 cm) within the regions accessible by endoscopic ultrasound in the pancreas, peripancreatic area, liver, adrenal gland, kidney, mediastinum, lung, and gastrointestinal submucosa. Biopsy is necessary for the diagnosis of these lesions;
* Must be able to receive examinations in the research center;
* Must be able to sign the informed consent.

Exclusion Criteria:

* Hemoglobin ≤8.0 g/dL;
* Pregnant women;
* Coagulation disorders (PLT <50,000/mm3,INR > 1.5);
* Took anticoagulants such as aspirin, warfarin in the latest week;
* Acute pancreatitis in the past two weeks;
* inability to safely perform EUS-TA (eg, cardiorespiratory dysfunction, mental diseases, or drug addiction); refusal or inability to provide an informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The histological diagnostic yields | up to 15 months
  The investigators' primary outcome measure is to compare the histological diagnostic yields of 22G Adapt Aspiration FNB and FNA puncture needle (22G EchoTip Ultra Echo-3-22) to the solid pancreatic or nonpancreatic lesions compared to conventional FNA puncture needle(22G EchoTip Ultra Echo-3-22) for pancreatic and non-pancreatic solid lesions.

SECONDARY OUTCOMES:
the histological acquisition yields | up to 15 months
  Comparing the histological acquisition yields of 22G Adapt Aspiration (EUS-FNB) and Echo-3-22 (EUS-FNA) for solid space-occupying lesions.
the diagnostic yields of the first pass and the number of subsequent passes | up to 15 months
  Comparing the diagnostic yields of the first puncture needle and subsequent puncture needles of 22G Adapt Aspiration (EUS-FNB) and Echo-3-22 (EUS-FNA) for solid space-occupying lesions(EUS-FNA) for the number of first and subsequent puncture needles for solid space occupying lesions.
the cytological diagnosis yields | up to 15 months
  Comparing the cytological diagnostic yields of 22G Adapt Aspiration (EUS-FNB) and Echo-3-22 (EUS-FNA) for solid space-occupying lesions.
the complication yields | up to 15 months
  Comparing the complication rates during and after puncture between 22G Adapt Aspiration (EUS-FNB) and Echo-3-22.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China

REFERENCES:
- [Result] Gkolfakis P, Crino SF, Tziatzios G, Ramai D, Papaefthymiou A, Papanikolaou IS, Triantafyllou K, Arvanitakis M, Lisotti A, Fusaroli P, Mangiavillano B, Carrara S, Repici A, Hassan C, Facciorusso A. Comparative diagnostic performance of end-cutting fine-needle biopsy needles for EUS tissue sampling of solid pancreatic masses: a network meta-analysis. Gastrointest Endosc. 2022 Jun;95(6):1067-1077.e15. doi: 10.1016/j.gie.2022.01.019. Epub 2022 Feb 4. PMID 35124072
- [Result] van Riet PA, Erler NS, Bruno MJ, Cahen DL. Comparison of fine-needle aspiration and fine-needle biopsy devices for endoscopic ultrasound-guided sampling of solid lesions: a systemic review and meta-analysis. Endoscopy. 2021 Apr;53(4):411-423. doi: 10.1055/a-1206-5552. Epub 2020 Aug 6. PMID 32583392
- [Result] Cheng B, Zhang Y, Chen Q, Sun B, Deng Z, Shan H, Dou L, Wang J, Li Y, Yang X, Jiang T, Xu G, Wang G. Analysis of Fine-Needle Biopsy vs Fine-Needle Aspiration in Diagnosis of Pancreatic and Abdominal Masses: A Prospective, Multicenter, Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1314-1321. doi: 10.1016/j.cgh.2017.07.010. Epub 2017 Jul 19. PMID 28733257
- [Result] Pouw RE, Barret M, Biermann K, Bisschops R, Czako L, Gecse KB, de Hertogh G, Hucl T, Iacucci M, Jansen M, Rutter M, Savarino E, Spaander MCW, Schmidt PT, Vieth M, Dinis-Ribeiro M, van Hooft JE. Endoscopic tissue sampling - Part 1: Upper gastrointestinal and hepatopancreatobiliary tracts. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2021 Nov;53(11):1174-1188. doi: 10.1055/a-1611-5091. Epub 2021 Sep 17. PMID 34535035
- [Result] Itonaga M, Yasukawa S, Fukutake N, Ogura T, Asada M, Shimokawa T, Inatomi O, Nakai Y, Shiomi H, Nebiki H, Suzuki A, Kitagawa K, Asai S, Shimatani M, Sanuki T, Kurita A, Takenaka M, Yoshida M, Hoki N, Yasuda H, Maruyama H, Matsumoto H, Yanagisawa A, Kitano M. Comparison of 22-gauge standard and Franseen needles in EUS-guided tissue acquisition for diagnosing solid pancreatic lesions: a multicenter randomized controlled trial. Gastrointest Endosc. 2022 Jul;96(1):57-66.e2. doi: 10.1016/j.gie.2022.02.005. Epub 2022 Feb 11. PMID 35151711
- [Result] Ashat M, Klair JS, Rooney SL, Vishal SJ, Jensen C, Sahar N, Murali AR, El-Abiad R, Gerke H. Randomized controlled trial comparing the Franseen needle with the Fork-tip needle for EUS-guided fine-needle biopsy. Gastrointest Endosc. 2021 Jan;93(1):140-150.e2. doi: 10.1016/j.gie.2020.05.057. Epub 2020 Jun 9. PMID 32526235
- [Result] Kurita A, Yasukawa S, Zen Y, Yoshimura K, Ogura T, Ozawa E, Okabe Y, Asada M, Nebiki H, Shigekawa M, Ikeura T, Eguchi T, Maruyama H, Ueki T, Itonaga M, Hashimoto S, Shiomi H, Minami R, Hoki N, Takenaka M, Itokawa Y, Uza N, Hashigo S, Yasuda H, Takada R, Kamada H, Kawamoto H, Kawakami H, Moriyama I, Fujita K, Matsumoto H, Hanada K, Takemura T, Yazumi S. Comparison of a 22-gauge Franseen-tip needle with a 20-gauge forward-bevel needle for the diagnosis of type 1 autoimmune pancreatitis: a prospective, randomized, controlled, multicenter study (COMPAS study). Gastrointest Endosc. 2020 Feb;91(2):373-381.e2. doi: 10.1016/j.gie.2019.10.012. Epub 2019 Oct 22. PMID 31654634